CLINICAL TRIAL: NCT00323505
Title: A Phase II Trial Comparing the Quality of Life, Tolerability and Toxicity of PEG Intron With INTRON® A in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1871
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2006-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Interferon alpha-2

INTERVENTIONS:
Drug: Pegylated Interferon
Drug: Interferon-alpha2a

SUMMARY:
Multiple myeloma is a rare form of malignancy in which neoplastic plasma cells accumulate in the bone marrow. Most malignant plasma cells continue to produce immunoglobulin. The activity of multiple myeloma can therefore usually be monitored easily by serial measurement of the serum paraprotein levels. Except for a few patients who receive a donor bone marrow transplant, multiple myeloma remains incurable despite intensive chemotherapy. Its course is typically marked by periods of active disease alternating with increasingly shorter remissions.

Interferons are substances produced in human cells in response to a variety of stimuli, such as viral infection. When given to myeloma patients as part of maintenance treatment , interferon-alpha 2 b (INTRONA) has been shown to be of value in prolonging the periods of remission. Until now, INTRONA could only be given as injections under the skin, three times a week. Some patients experience flu-like symptoms with each injection, particularly early on during maintenance therapy. This, as well as the chronic fatigue and even depression that INTRONA can induce may considerably reduce the quality of life of myeloma patients on interferon, so much so that sometimes this useful adjunct to chemotherapy for myeloma has to be stopped.

Recently, a new preparation of interferon namely pegylated interferon (PEG Intron) has become available. It has the advantage of being broken down much more slowly by the body and therefore only needs to be given once a week. This minimises the swings in blood interferon levels that may be responsible for some of the interferon side effects. The safety and superior tolerability of PEG Intron has already been demonstrated in patients with hepatitis C for which it now carries a licence, but not in myeloma patients. Here, we propose to study whether the quality of life and side effect profile of myeloma patients on PEG Intron is better compared to that of Intron®A.

In the main study, consenting eligible myeloma patients who are well and have been established on INTRONA maintenance therapy for at least six weeks will be randomly allocated to receive PEG Intron for three months followed by INTRONA for 3 months, or to continue with INTRONA for 3 months followed by PEG Intron for 3 months. All patients will be monitored regularly for any side effects and will be asked to fill in a quality of life questionnaire at the beginning (i.e. before receiving the first randomised treatment) and at the end of each study period (i.e. at 3 and 6 months). Initially, we are aiming at enrolling 60 patients into this part of the study.

In a smaller sub-study involving only 14 patients initially, we are proposing to investigate whether myeloma patients who need to be taken off Intron®A because of its side effects can tolerate PEG Intron more easily. Should their tolerance of PEG Intron also be poor we would stop the interferon maintenance therapy altogether. However, should PEG Intron be found to be acceptable to them, we intend to switch these patients back to the standard treatment at the end of six weeks treatment with PEG Intron to assess whether they have become more tolerant of Intron®A in the intervening period. Patients will again be monitored carefully for any side effects and will be asked to fill in three quality of life questionnaires (at 0, 6 and 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Patients  18 years of age with a definite diagnosis of multiple myeloma.
2. Patients have been on a steady dose of INTRON®A for at least 6 weeks and have tolerated it (randomized study only), or patients who within six weeks of starting INTRON®A become intolerant (tolerability sub-study only)
3. Informed consent obtained

Exclusion Criteria:

- a) Patients with refractory Multiple Myeloma. b) Treatment with any investigational drug within 30 days of entry to this protocol.

c) Subjects who are pregnant, nursing, or of reproductive potential and who are not practising an effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Ray Powles, FRCP, FRCpath, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS trust, Sutton, Surrey, United Kingdom